CLINICAL TRIAL: NCT06408467
Title: Monitoring of Non-Surgical Treatment of Peri-implantitis, Traditional Measurement Methods and aMMP-8 Test Technology-Cross Sectional Study
Brief Title: Monitoring of Non-Surgical Treatment of Peri-implantitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lahanna oy (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Lahanna
Record Dates: First submitted 2024-05-02; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Peri-implant Mucositis; Peri-Implantitis
Keywords: peri-implant treatment; aMMP-8; non-surgical treatment
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The effect and monitoring of maintenance therapy for peri-implantitis (Experimental)
  Interventions: Other: aMMP-8 diagnostic test

INTERVENTIONS:
Other: aMMP-8 diagnostic test — 40 patients

SUMMARY:
This study aimed to investigate the response to non-surgical treatment of peri-implantitis diseases during the maintenance phase. The patients underwent non-surgical implant maintenance treatment, and the success of the treatment was measured again after 30 days using the same criteria and methods.

DETAILED DESCRIPTION:
For 40 patients, the aMMP-8 test was performed on the buccal gingival pocket of the implant teeth, gingival bleeding (BOP), implant pocket depth (PPD), and a periapical x-ray to measure radiologic bone level (RBL) were taken.

ELIGIBILITY:
Inclusion Criteria:

* implant patients arriving for a maintenance visit at a dental clinic
* a diagnosis of peri-implant healthy, peri-implant mucositis, or peri-implantitis by a dentist
* a written informed consent.

Exclusion Criteria

* Smoking
* age under 25
* antibiotic treatment within six months
* the maintenance treatment had been completed within 6 months.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
the result of the participants who were measured aMMP-8 | 1 month
  Measure aMMP-8-level ng/ml
the result of the participants who were measured BOP | 1 month
  measure bleeding on probing in PISF
the result of the participants who were measured PPD | 1 month
  measure peri-implant pocket depth

CONTACTS AND LOCATIONS:
Overall Officials: Timo Sorsa, Professor, Study Director — University of Helsinki
Locations (1):
- University of Helsinki, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available after the research
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting in June 2025 and end of January 2026
Access Criteria: information can be shared with an email request to share IPD and other support information. Requests are reviewed with the research team.

REFERENCES:
- [Result] Lindhe J, Meyle J; Group D of European Workshop on Periodontology. Peri-implant diseases: Consensus Report of the Sixth European Workshop on Periodontology. J Clin Periodontol. 2008 Sep;35(8 Suppl):282-5. doi: 10.1111/j.1600-051X.2008.01283.x. PMID 18724855
- [Result] Figuero E, Graziani F, Sanz I, Herrera D, Sanz M. Management of peri-implant mucositis and peri-implantitis. Periodontol 2000. 2014 Oct;66(1):255-73. doi: 10.1111/prd.12049. PMID 25123773
- [Result] Lahteenmaki H, Umeizudike KA, Heikkinen AM, Raisanen IT, Rathnayake N, Johannsen G, Tervahartiala T, Nwhator SO, Sorsa T. aMMP-8 Point-of-Care/Chairside Oral Fluid Technology as a Rapid, Non-Invasive Tool for Periodontitis and Peri-Implantitis Screening in a Medical Care Setting. Diagnostics (Basel). 2020 Aug 5;10(8):562. doi: 10.3390/diagnostics10080562. PMID 32764436
- [Result] Alassy H, Parachuru P, Wolff L. Peri-Implantitis Diagnosis and Prognosis Using Biomarkers in Peri-Implant Crevicular Fluid: A Narrative Review. Diagnostics (Basel). 2019 Dec 7;9(4):214. doi: 10.3390/diagnostics9040214. PMID 31817894
- [Derived] Lahteenmaki H, Raisanen IT, Tervahartiala T, Parnanen P, Patila T, Sorsa T. Monitoring of Nonsurgical Treatment of Peri-Implantitis Traditional Measurement Methods and aMMP-8 Test Technology: A Pilot Study. Int J Dent. 2025 Nov 27;2025:6681032. doi: 10.1155/ijod/6681032. eCollection 2025. PMID 41358008